CLINICAL TRIAL: NCT00668694
Title: Effect of Psychosocial Stimulation on Development of Iron-deficient Anemic Infants: A Randomized Controlled Trial
Brief Title: Iron Deficiency Anemia and Psychosocial Stimulation
Acronym: IDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Dhaka, Bangladesh (Other); Institute of Child Health (Other); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-040
Record Dates: First submitted 2008-04-27; First posted 2008-04-29 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2008-04

CONDITIONS: Iron Deficiency Anemia
Keywords: Psychosocial stimulation in addition to iron supplementation will improve mental and psychomotor development, language, behavior and growth of IDA infants.; With the addition of stimulation IDA infants will catch up to the non-anemic infants.
MeSH Terms: conditions — Anemia, Iron-Deficiency; Language; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (No Intervention): Anemia without stimulation.
- 2 (Experimental): Anemia with stimulation
  Interventions: Behavioral: Stimulation
- 3 (No Intervention): Non-anemic group: Hb >80-109 g/L ferritin levels >12 μg/L and TfR <6 will be enrolled without stimulation
- 4 (No Intervention): Non-anemic group: Hb >80-109 g/L ferritin levels >12 μg/L and TfR <6 will be enrolled with stimulation

INTERVENTIONS:
Behavioral: Stimulation — Stimulation given to the child by mother
  Arms: 2

SUMMARY:
In developing countries, poor nutrition, high morbidity, poverty, poor parental education and stimulation in the home, all detrimentally affect children's development. These conditions frequently occur together increasing the risk of poor development. Iron deficiency anemia (IDA) affects large numbers of young children and is associated with poor child development. There is some question as to whether infants with IDA can catch up in mental development to non-IDA infants. We plan to examine the effect of psychosocial stimulation on IDA children's growth and development using a randomized controlled trial and compare them with non-anemic children. The study will be located in poor villages accessible to Dhaka. Villages will be randomized to either receive psychosocial stimulation or none. Children, aged 6-12 months, with IDA (hemoglobin (Hb) 80.0-109g/L, ferritin<12μg/L & Transferrin Recepter (TfR) >7) (n=212) or without anemia (Hb>109g/L, ferritin>12μg/L, C-reactive protein (CRP) <5 & TfR<7) (n=212) will be identified in those villages. Intervention will include weekly home visits for 9 months by a play leader, who will demonstrate play with home made toys and teach the mothers about child development. All IDA children will be given 30 mg ferrous-sulphate daily for 9 months. At the beginning and end of the study, the following measurements will be made: Bayley Scales of Infant Development (mental and motor indices), Wolke's behavior ratings, Hb, serum ferritin, CRP, Transferrin receptor, anthropometry, home stimulation, and mothers' knowledge and practices of child development. Stool microscopy, maternal-urinary iodine (as a proxy to assess children's iodine status), dietary history, child rearing practices (parenting) of mothers, perinatal history and socioeconomic conditions will be assessed at the beginning and children's language development at the end. Depending on availability of funds serum TSH will also be measured in children to exclude iodine deficiency. We will also measure mothers' nutritional and mental status to assess its relationship with children's development. The treatment effect will be examined by intention to treat analysis using multiple regression of the outcome variables controlling for initial measures and multilevel analysis will be conducted to control for differences at village level. The findings of this project will have implications both for international and national policies on early childhood development programs for IDA children.

DETAILED DESCRIPTION:
In developing countries, millions of young children have developmental deficits due to poor nutrition, lack of a stimulating environment, and poverty. In Bangladesh, where poor nutrition, poverty and poor parental education are highly prevalent, the implications are serious not only for the individuals' future but also for national development.

Iron deficiency and child development There is increasing evidence that iron deficiency anemia detrimentally affects children's development (Grantham-McGregor and Ani 2001). Many cross sectional studies have shown that iron deficiency is associated with poor psychomotor development and behavioral deficits in young children, and poor cognition and school achievement in school-aged children. Furthermore, longitudinal studies have observed that children who are anemic in the first 3 years of life continue to have poorer cognition, school achievement and psychosocial well being than children who were not anemic (Grantham-McGregor and Ani 2001). However, anemia is associated with many adverse social and economic family circumstances (Lozoff et al. 1991;de Andraca et al. 1990), which may adversely affect children's development.

Anemic children who were treated with iron, failed to catch up with non-anemic children in developmental levels in several studies (e.g. Walter et al. 1989;Lozoff et al. 1987;Lozoff et al. 1996). A few randomized, controlled trials of iron treatment have been conducted with anemic young children (Stoltzfus et al. 2001;Idjarinata and Pollitt 1993;Aukett et al. 1986;Friel et al, 2001). In two of the trials, anemic children under four (Stoltzfus et al. 2001) or two years (Idjarinata and Pollitt 1993) achieved better development from iron supplementation. One of these studies in Indonesia involved only 25 treated anemic children (Idjarinata and Pollitt 1993). The other study was in Zanzibar and included many children with malaria and some severely anemic children (Stoltzfus et al. 2001) and only children with Hb <80g/L showed significant benefits in motor development but improvement in language milestones occurred in children with all levels of Hb. Two other randomized trials failed to show clear benefits (Aukett et al. 1986;Friel et al, 2001). One of them (Aukett et al. 1986) used an insensitive screening test to measure developmental outcomes and the other (Friel et al, 2001) compared the effect of low and high iron formula on the development of low birth weight children and no benefit was found in the high iron group. The high iron children actually had more respiratory infections.

A recent meta-analysis of randomised trials (Sachdev et al, 2005) found that while there is evidence that older anemic children benefit from iron in cognition there is no convincing evidence from children under 27 months. However, three more recent randomized trials of iron supplementation were not included (Black et al, 2004; Lind et al, 2004, Freil et al 2003). One in Bangladesh (Black et al, 2004) found a non significant benefit to motor development from iron alone however the power of the study was extremely limited and the group receiving iron and zinc benefited in motor development. Both the Indonesian (Lind et al, 2004) and Canadian studies (Freil et al 2003) found benefits from iron treatment to infants' motor development but not to mental development. It has been suggested that the poor level of mental development found in IDA infants may be irreversible in some circumstances (Lozoff et al 2000).

Stimulation and child development Iron deficient children show less activity, more apathy and are less likely to explore their environment than iron replete children and thus acquire skills only slowly (Grantham-McGregor and Ani 2001). One reason for the failure of some anemic children to catch up in mental development to non-anemic children following treatment may be that they have missed opportunities to explore their environment. Thus, they may require extra play experiences to catch up in development. In addition, many anemic children come from homes with low levels of stimulation and other psychosocial disadvantages (Grantham-McGregor and Ani 2001), which may exacerbate their poor level of development.

In previous studies in poor populations, it has been shown that teaching mothers how to play with their children and be responsive to them improves the children's development (WHO 1999). It is clear that in order to reach their developmental potential, disadvantaged children require not only good health and nutrition but also supportive and caring environments. In Jamaica (Grantham-McGregor et al. 1991), stunted children needed extra stimulation as well as food supplementation to catch up with non-stunted children. We therefore plan to examine the benefits of adding psychosocial stimulation to iron treatment on IDA infants motor and mental development and determine if they catch up to non-anemic infants.

Situation in Bangladesh The nutritional status of Bangladeshi children is extremely poor. Low birth weight is estimated to occur in 36% of births. It is estimated that among children under 5 years the prevalence of stunting (height-for-age <-2 z scores) is 43% and wasting (weight-for-height <-2 z scores) is 13% (UNICEF 2006). Iron deficiency anemia is a major public health problem in young children. A national rural survey found that 52.7% of children aged 6 to 59 months were anemic (Hb <110g/L). However, the prevalence of anemia was 78% among children 6-11 months of age and 64% among children 12- 23 months of age (IPHN/HKI 1999). A review of studies of prevalence of anemia in Bangladesh (Ahmed 2000) found levels ranging from 81 to 49% with a suggestion of rural children having higher levels of anemia than urban children in small studies. However, severe anemia (Hb < 70g/L) was rare.

The main etiology of anemia in young children in Bangladesh is reported to be poor dietary iron intake especially during the period of rapid growth (Ahmed 2000). Vitamin A deficiency is common and may contribute to anemia (Ahmed et al. 2001). However, in Bangladesh there is a government policy of supplementing children under 5 years with vitamin A every 6 months and coverage is estimated to be good at 87% (UNICEF 2006). A national survey in 1995-6 (Jahan and Hossain 1998) found that the diets of children aged one to three years have marked deficits in energy, protein and iron. Approximately 60% of iron intake came from cereal. It is clear that poor iron intake is a major contributor to iron deficiency in this population. Low birth weight is also highly prevalent and low iron stores from birth are likely to be another important contributor to iron status.

A representative survey of 14 rural districts (7,764 people of 0-60 years of age) found that anemia was associated with large families, poor sanitation and socioeconomic status, poor nutritional status and parasitic infection (Husain et al. 1997). Anemic children are therefore likely to be exposed to several risk factors associated with poverty that may detrimentally affect their development.

Iodine deficiency was endemic in Bangladesh and national Iodine Deficiency Disorder (IDD) survey in 1993 found 47.1% of population suffered from some form of goiter and about 69% of people were biochemically iodine deficient (Yusuf et al. 1993). Following this survey, salt iodination program was started in 1993, which has improved the iodine status of the people in the country. In 1998 a nationwide survey found that 77% of households (in the whole country except in Cox's Bazar district) consumed iodized salt (BBS 1998). According to the UNICEF's report 70% of all households in Bangladesh consume iodized salt (UNICEF 2006). We will therefore assess whether iodine deficiency is a problem in the study population and if so, we will advice the families to use iodized salt.

In addition most Bangladeshi mothers suffer from poor nutrition (The March of Dimes, 2002), anemia (Stallkamp et al. 2006), low education (Unicef 2006), and some are also depressed (Hamadani, personal communication). Maternal nutritional (Perez et al. 2005) and mental status (Black et al. 2007) has been found to affect children's development.

ELIGIBILITY:
Inclusion Criteria:

* All children will be aged 6 to 24 months, living in the defined rural area and have parental consent to join the study

Exclusion Criteria:

* The following children will be excluded:

  * those with multiple births
  * congenital abnormalities
  * Bayley scores <55
  * Hb<80 g/L or severe wasting (weight for height <-3 z score)
* Children with severe wasting or Hb<80 g/L will be referred to the Thana Health Complex for treatment.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 434 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Mental and motor development. | 9 months

SECONDARY OUTCOMES:
Anthropometry | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Background] Tofail F, Hamadani JD, Mehrin F, Ridout DA, Huda SN, Grantham-McGregor SM. Psychosocial stimulation benefits development in nonanemic children but not in anemic, iron-deficient children. J Nutr. 2013 Jun;143(6):885-93. doi: 10.3945/jn.112.160473. Epub 2013 Apr 24. PMID 23616511